CLINICAL TRIAL: NCT04837729
Title: The Effect of Acupressure Applied to Menopausal Women on Menopausal Symptoms and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ahu AKSOY, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 701
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Menopausal Symptom; Quality of Life
Keywords: Acupressure; Menopause; Menopausal symptoms; Quality of life; Nursing
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (acupressure) group (Experimental): Acupressure (complementary and integrative medicine method) Acupressure will be applied individually to the experimental group for 20-25 minutes three times a week for four weeks. Data collection forms will be applied 3 times in total, before the intervention, in the second and the fourth week.
  Interventions: Other: Acupressure
- Control group (No Intervention): No intervention will be made to women in the control group. However, data collection forms will be applied 3 times in total, before the intervention, in the second and the fourth week.

INTERVENTIONS:
Other: Acupressure — acupressure is a non-pharmacological method originating from traditional Chinese medicine. According to the National Cancer Institute, acupressure is defined as pressure / massage applied to certain parts of the body to control symptoms such as pain or nausea. The main purpose of acupressure is to stimulate the regions associated with the specific organ by applying pressure with energy channels called meridians.
  Arms: Experimental (acupressure) group

SUMMARY:
In this randomized controlled study, it was aimed to determine the effect of acupressure on menopausal symptoms and quality of life and the relationship between menopausal symptoms and quality of life. Three different hypothesis teams have been established for the study. These; H0: There is no significant difference between the menopause rating scores of the women in the study group in which acupressure was applied and the control group without acupressure.

H1: There is a significant difference between the menopause rating scores of the women in the study group in which acupressure was applied and the control group without acupressure.

H0: There is no significant difference between the quality of life scores of the women in the study group in which acupressure was applied and the control group without acupressure.

H1: There is a significant difference between the quality of life scores of the women in the study group in which acupressure was applied and the control group without acupressure.

H0: There is no relationship between menopause rating scores and quality of life scores of women in the study group in which acupressure was applied and in the control group without acupressure.

H1: There is a relationship between menopause rating scores and quality of life scores of women in the study group in which acupressure was applied and in the control group without acupressure.

DETAILED DESCRIPTION:
Parallel to the increase in life expectancy by years, the population of women living in the post-menopausal period is also increasing. In order to have a healthy menopause, which is an important part of women's life, it is thought that the acupressure without health risks by women may be effective in reducing the symptoms of menopause experienced by women and quality of life. In line with this information, it was aimed to determine the effect of acupressure on menopausal symptoms and quality of life and the relationship between menopausal symptoms and quality of life. The study will be carried out with menopausal women between the ages of 40-60 in Mersin province in Turkey. Therefore, in the study, 46 women in the menopausal period between the ages of 40-60 will be randomly assigned to acupressure and control groups. The study group (n = 23) will be applied to the determined points in a certain order. Sequence of application Large intestine 4th point (LI 4), Heart 7th point (HT 7), Triple warmer point 23 (TE 23), Stomach 36th point (ST 36), Spleen 6th point (SP 6) and Liver The 3rd point is (LV 3). Acupressure application for 20-25 minutes three times a week for four weeks will be applied individually to the study group. No intervention will be made to the control group for a period of four weeks. The primary expected outcome of the research is the effect of acupressure on menopausal symptoms of menopausal women. The second expected result of the study is to determine the effect of acupressure on quality of life. Results will be applied three times in total, before the study and control application, two weeks and 4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in research,
* Can read and write in Turkish,
* Open to communication,
* Those who are between the ages of 40-60 and do not experience menstruation for at least one year,
* Experiencing at least one or more of the menopausal symptoms,
* Do not use medication for the treatment of menopausal symptoms,
* No chronic disease,
* Body mass index <30 kg / m2,
* Not applying regular acupressure,
* Those who have not surgically entered menopause,
* Women without psychiatric problems

Exclusion Criteria:

* - who do not agree to participate in the research,
* Can't read and write Turkish,
* Communication is not possible,
* Those who are younger than 40, older than 60, have experienced menstruation for at least one year,
* Do not experience the symptoms of menopause,
* Using medication for the treatment of menopausal symptoms,
* Chronic illness,
* Body mass index ≥30 kg / m2,
* Regular acupressure is applied,
* Surgically in menopause,
* Women with psychiatric problems

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 40-60 who are in menopause
Enrollment: 61 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale | change from before intervention, 2nd and 4th week of intervention
  It was developed in German by Schneider et al. In 1992 to measure the severity of menopausal symptoms and was adapted to English in 1996. MRT was adapted to Turkish by Gürkan in our country in 2005. There are "0 = None", "1 = Mild", "2 = Moderate", "3 = Severe" and "4 = Very severe" options for each item in the Likert-type scale consisting of 11 items including menopausal complaints. The total score of the scale is calculated based on the scores given for each item. The lowest score that can be obtained from the scale is 0, the highest score is 44.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF) | change from before intervention, 2nd and 4th week of intervention
  Life of quality will be evaluated by using the WHOQOL-BREF-TR. This scale consists of 27 questions. There are a total of five areas in the scale: physical, mental, social, environmental and national environmental areas. Each area is evaluated within itself. The domain score is calculated with the score it gets from the questions that determine it. Field scores are evaluated between 4-20. Increasing score indicates goodness. Cronbach's alpha internal consistency coefficients of the scale; 0.83 in the physical area, 0.66 in the spiritual area, 0.53 in the social area, 0.73 in the environmental area and 0.73 in the national environmental area.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu VEFİKULUÇAY YILMAZ, Dr., Study Director — Mersin University Nursing Faculty
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kao YH, Huang YC, Chung UL, Hsu WN, Tang YT, Liao YH. Comparisons for Effectiveness of Aromatherapy and Acupressure Massage on Quality of Life in Career Women: A Randomized Controlled Trial. J Altern Complement Med. 2017 Jun;23(6):451-460. doi: 10.1089/acm.2016.0403. Epub 2017 May 15. PMID 28504569
- [Background] Ahmadinezhad M, Kargar M, Vizeshfar F, Hadianfard MJ. Comparison of the Effect of Acupressure and Pilates-Based Exercises on Sleep Quality of Postmenopausal Women: A Randomized Controlled Trial. Iran J Nurs Midwifery Res. 2017 Mar-Apr;22(2):140-146. doi: 10.4103/1735-9066.205954. PMID 28584553
- See also: Effect of acupressure on early complications of menopause in women referring to selected health care centers — https://www.ijnmrjournal.net/crossrefCitation.asp?doi=10.4103/1735-9066.208165